CLINICAL TRIAL: NCT02422485
Title: A 6 Month, Open-Label, Pilot Futility Clinical Trial of Oral Salsalate for Progressive Supranuclear Palsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adam Boxer (Other)
Responsible Party: Sponsor-Investigator, Adam Boxer, MD, PhD, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Salsalate PSP
Record Dates: First submitted 2015-04-09; First posted 2015-04-21 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Progressive Supranuclear Palsy
Keywords: Salsalate
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — salicylsalicylic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Salsalate (Experimental): All participants will be administered 2,250 mg daily [1,500 mg every day before noon (every AM) and 750 mg every night at bedtime (every HS)] for 6 months.
  Interventions: Drug: Salsalate

INTERVENTIONS:
Drug: Salsalate — Salsalate is a non-acetylated dimer of salicylic acid, and is classified as a NSAID. The chemical name of salsalate is 2-hydroxy-benzoic acid, 2-carboxyphenyl ester. Salsalate has a molecular weight (MW) of 258.226 Da and a molecular formula of C14H10O5.

SUMMARY:
This is a multi-center, open label, pilot futility clinical trial of the safety, tolerability, pharmacodynamics and preliminary efficacy of oral salsalate in up to 10 patients with PSP.

DETAILED DESCRIPTION:
This is a multi-center, open label, pilot futility clinical trial of the safety, tolerability, pharmacodynamics and preliminary efficacy of oral salsalate in up to 10 patients with PSP. All participants will be administered 2,250 mg daily [1,500 mg every day before noon (every AM) and 750 mg every night at bedtime (every HS)] for 6 months.

If ≥3 patients experience drug limiting toxicity (DLT), as defined below, the study will be terminated.

A DLT is defined as: 1) any Grade 3 or higher adverse event (AE) per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) for which there is reasonable possibility that salsalate caused the event, 2) any Grade 2 AE in the CTCAE system organ class of nervous system disorders that is considered clinically significant and for which there is reasonable possibility that salsalate caused the event, or 3) any Grade 2 or higher treatment-related adverse events during administration that do not resolve promptly with supportive treatment.

An interim futility analysis will be performed after five subjects have completed 6 months of study drug treatment. If the criteria listed in the Statistical Methods section of this synopsis are met, an additional 5 subjects will be enrolled in the trial. If not, the trial will be terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Meets National Institute of Neurological Disorders and Stroke - Society for Progressive Supranuclear Palsy (NINDS-SPSP) probable or possible PSP criteria,(Litvan 1996a) as modified from the AL-108-231 trial.(Boxer 2014)
2. Aged 50-85
3. Agrees to 3 magnetic resonance imaging (MRI) or subject to investigator's discretion
4. MRI at screening is consistent with PSP (≤4 microhemorrhages and no large strokes or severe white matter disease)
5. Mini-Mental State Examination (MMSE) score 14-30
6. Stable medications for 2 months prior to screening, including FDA approved Alzheimer's disease (AD) medications and Parkinson's disease medications
7. Availability of a study partner who knows the patient well and is willing to accompany the patient to all trial visits and to participate in questionnaires
8. Agrees to 2 lumbar punctures for cerebrospinal fluid (CSF) examination
9. Signed and dated written informed consent obtained from the subject and subject's caregiver in accordance with local IRB regulations
10. Males and all WCBP agree to abstain from sex or use an adequate method of contraception for the duration of the study and for 30 days after the last dose of study drug.

    * Adequate contraceptive methods include those with a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as complete abstinence from sexual intercourse with a potentially fertile partner, and some double barrier methods condom with spermicide) in conjunction with use by the partner of an intrauterine device (IUD), diaphragm with spermicide, oral contraceptives, birth control patch or vaginal ring, oral, or injectable or implanted contraceptives.
    * For this study, a woman who has been surgically sterilized or who has been in a state of amenorrhea for more than two years will be deemed not to be of childbearing potential;

Exclusion Criteria:

1. Meets National Institute on Aging-Alzheimer's Association Workgroups criteria for probable AD (McKhann et al. 2011);
2. Any medical condition other than PSP that could account for cognitive deficits (e.g., active seizure disorder, stroke, vascular dementia);
3. A prominent and sustained response to levodopa therapy;
4. History of significant cardiovascular, hematologic, renal, or hepatic disease (or laboratory evidence thereof);
5. History of hypertension (repeated elevations in blood pressure exceeding 180 mm Hg systolic or 100 mm Hg diastolic; medical intervention indicated);
6. History of severe gastrointestinal bleed, or gastric or peptic ulcers;
7. History of aspirin triad (i.e., aspirin allergy, nasal polyps and asthma) or asthma;
8. History of major psychiatric illness or untreated depression;
9. Neutrophil count <1,500/mm3, platelets <100,000/mm3, serum creatinine >1.5 x upper limit of normal (ULN), total bilirubin >1.5 x ULN, alanine aminotransferase (ALT) >3 x ULN, aspartate aminotransferase (AST) >3 x ULN, or INR >1.2 at Screening evaluations;
10. Evidence of any clinically significant findings on Screening or baseline evaluations which, in the opinion of the Investigator would pose a safety risk or interfere with appropriate interpretation of study data;
11. Current or recent history (within four weeks prior to Screening) of a clinically significant bacterial, fungal, or mycobacterial infection;
12. Current clinically significant viral infection. Subjects with chicken pox, influenza, or flu symptoms are not eligible;
13. Major surgery within four weeks prior to Screening;
14. Any contraindication to or unable to tolerate lumbar puncture at Screening, including use of anti-coagulant medications such as warfarin. Daily administration of 81 mg aspirin will be allowed as long as the dose is stable for 30 days prior to Screening;
15. Treatment with another investigational drug or participation in another interventional clinical trial within 3 months of Screening;
16. Chronic use of other NSAIDs or salicylates for any reason, except for daily baby aspirin (81 mg);
17. Concurrent treatment with thiazides or loop diuretics;
18. Concurrent use of oral corticosteroids or angiotensin-converting enzyme (ACE) inhibitors;
19. Treatment with any human blood product, including intravenous immunoglobulin, during the 6 months prior to Screening or during the trial;
20. Known hypersensitivity to the inactive ingredients in the study drug;
21. Pregnant or lactating;
22. Positive pregnancy test at Screening or Baseline (Day 1);
23. Cancer within 5 years of Screening, except for non-metastatic skin cancer or nonmetastatic prostate cancer not expected to cause significant morbidity or mortality within one year of Baseline.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing drug limiting toxicity (DLT), | 6 months
  defined as: 1) any Grade 3 or higher adverse event (AE) per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) for which there is reasonable possibility that salsalate caused the event, 2) any Grade 2 AE in the CTCAE system organ class of nervous system disorders that is considered clinically significant and for which there is reasonable possibility that salsalate caused the event, or 3) any Grade 2 or higher treatment-related adverse events during administration that do not resolve promptly with supportive treatment.

SECONDARY OUTCOMES:
Changes in motor function | 6 months
  Motor function as measured by Progressive Supranuclear Palsy Rating Scale (PSPRS) comprising 28 items in six categories: daily activities (by history), behavior, bulbar, ocular motor, limb motor and gait/midline The available total score ranges from 0 to 100; lower scores reflect better outcome.
Changes in cognition | 6 months
  Cognitive function as measured by Progressive Supranuclear Palsy Rating Scale (PSPRS) comprising 28 items in six categories: daily activities (by history), behavior, bulbar, ocular motor, limb motor and gait/midline The available total score ranges from 0 to 100; lower scores reflect better outcome.
Changes in activities of daily living | 6 months
  Activities of daily living as measured by Progressive Supranuclear Palsy Rating Scale (PSPRS) comprising 28 items in six categories: daily activities (by history), behavior, bulbar, ocular motor, limb motor and gait/midline The available total score ranges from 0 to 100; lower scores reflect better outcome.
Changes in behavior | 6 months
  Behavior as measured by Progressive Supranuclear Palsy Rating Scale (PSPRS) comprising 28 items in six categories: daily activities (by history), behavior, bulbar, ocular motor, limb motor and gait/midline The available total score ranges from 0 to 100; lower scores reflect better outcome.

OTHER OUTCOMES:
Changes in concentration of cerebrospinal fluid (CSF) biomarkers | 6 months
  Changes in the concentrations of cerebrospinal fluid (CSF) biomarkers
Changes in brain volume | 6 months
  Changes in brain volume [T1-weighted volumetric magnetic resonance imaging (vMRI)], brain network functional and structural connectivity and perfusion [resting state functional magnetic resonance imaging (rsfMRI), diffusion tensor imaging (DTI), and arterial spin labeling (ASL) perfusion magnetic resonance imaging (MRI)]
Changes in motor function, cognition, activities of daily living, and behavior | 6 months
  Motor function, cognition, activities of daily living, and behavior as measured by Schwab and England Activities of Daily Living scale (SEADL), PSP-Quality of Life. Scores range from one hundred percent, which indicates a completely independent individual, and zero percent, which indicates an individual in who is no longer functioning.
Changes in saccade eye movements | 6 months
  To explore the effects of 2,250 mg daily salsalate on changes in saccade latency, velocity, and amplitude [infrared oculometry] from Screening to end of month 3 and end of month 6 compared to historical data;
Changes in sleep and activity levels | 6 months
  Changes in actigraphic measures

CONTACTS AND LOCATIONS:
Overall Officials: Adam Boxer, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - OHSU Parkinson Center & Movement Disorder Program, Portland, Oregon

REFERENCES:
- [Background] Bensimon G, Ludolph A, Agid Y, Vidailhet M, Payan C, Leigh PN; NNIPPS Study Group. Riluzole treatment, survival and diagnostic criteria in Parkinson plus disorders: the NNIPPS study. Brain. 2009 Jan;132(Pt 1):156-71. doi: 10.1093/brain/awn291. Epub 2008 Nov 23. PMID 19029129
- [Background] Boxer AL, Lang AE, Grossman M, Knopman DS, Miller BL, Schneider LS, Doody RS, Lees A, Golbe LI, Williams DR, Corvol JC, Ludolph A, Burn D, Lorenzl S, Litvan I, Roberson ED, Hoglinger GU, Koestler M, Jack CR Jr, Van Deerlin V, Randolph C, Lobach IV, Heuer HW, Gozes I, Parker L, Whitaker S, Hirman J, Stewart AJ, Gold M, Morimoto BH; AL-108-231 Investigators. Davunetide in patients with progressive supranuclear palsy: a randomised, double-blind, placebo-controlled phase 2/3 trial. Lancet Neurol. 2014 Jul;13(7):676-85. doi: 10.1016/S1474-4422(14)70088-2. Epub 2014 May 27. PMID 24873720
- [Background] Breen DP, Vuono R, Nawarathna U, Fisher K, Shneerson JM, Reddy AB, Barker RA. Sleep and circadian rhythm regulation in early Parkinson disease. JAMA Neurol. 2014 May;71(5):589-595. doi: 10.1001/jamaneurol.2014.65. PMID 24687146
- [Background] Brunden KR, Trojanowski JQ, Lee VM. Advances in tau-focused drug discovery for Alzheimer's disease and related tauopathies. Nat Rev Drug Discov. 2009 Oct;8(10):783-93. doi: 10.1038/nrd2959. PMID 19794442
- [Background] Cohen TJ, Guo JL, Hurtado DE, Kwong LK, Mills IP, Trojanowski JQ, Lee VM. The acetylation of tau inhibits its function and promotes pathological tau aggregation. Nat Commun. 2011;2:252. doi: 10.1038/ncomms1255. PMID 21427723
- [Background] Dugbartey AT, Townes BD, Mahurin RK. Equivalence of the Color Trails Test and Trail Making Test in nonnative English-speakers. Arch Clin Neuropsychol. 2000 Jul;15(5):425-31. PMID 14590218
- [Background] Fagan AM, Shaw LM, Xiong C, Vanderstichele H, Mintun MA, Trojanowski JQ, Coart E, Morris JC, Holtzman DM. Comparison of analytical platforms for cerebrospinal fluid measures of beta-amyloid 1-42, total tau, and p-tau181 for identifying Alzheimer disease amyloid plaque pathology. Arch Neurol. 2011 Sep;68(9):1137-44. doi: 10.1001/archneurol.2011.105. Epub 2011 May 9. PMID 21555603
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Gardner RC, Boxer AL, Trujillo A, Mirsky JB, Guo CC, Gennatas ED, Heuer HW, Fine E, Zhou J, Kramer JH, Miller BL, Seeley WW. Intrinsic connectivity network disruption in progressive supranuclear palsy. Ann Neurol. 2013 May;73(5):603-16. doi: 10.1002/ana.23844. Epub 2013 Mar 27. PMID 23536287
- [Background] Golbe LI, Ohman-Strickland PA. A clinical rating scale for progressive supranuclear palsy. Brain. 2007 Jun;130(Pt 6):1552-65. doi: 10.1093/brain/awm032. Epub 2007 Apr 2. PMID 17405767
- [Background] Golbe LI, Davis PH, Schoenberg BS, Duvoisin RC. Prevalence and natural history of progressive supranuclear palsy. Neurology. 1988 Jul;38(7):1031-4. doi: 10.1212/wnl.38.7.1031. PMID 3386818
- [Background] Goldfine AB, Fonseca V, Jablonski KA, Chen YD, Tipton L, Staten MA, Shoelson SE; Targeting Inflammation Using Salsalate in Type 2 Diabetes Study Team. Salicylate (salsalate) in patients with type 2 diabetes: a randomized trial. Ann Intern Med. 2013 Jul 2;159(1):1-12. doi: 10.7326/0003-4819-159-1-201307020-00003. PMID 23817699
- [Background] Knopman DS, Kramer JH, Boeve BF, Caselli RJ, Graff-Radford NR, Mendez MF, Miller BL, Mercaldo N. Development of methodology for conducting clinical trials in frontotemporal lobar degeneration. Brain. 2008 Nov;131(Pt 11):2957-68. doi: 10.1093/brain/awn234. Epub 2008 Oct 1. PMID 18829698
- [Background] Litvan I, Agid Y, Calne D, Campbell G, Dubois B, Duvoisin RC, Goetz CG, Golbe LI, Grafman J, Growdon JH, Hallett M, Jankovic J, Quinn NP, Tolosa E, Zee DS. Clinical research criteria for the diagnosis of progressive supranuclear palsy (Steele-Richardson-Olszewski syndrome): report of the NINDS-SPSP international workshop. Neurology. 1996 Jul;47(1):1-9. doi: 10.1212/wnl.47.1.1. PMID 8710059
- [Background] Litvan I, Agid Y, Jankovic J, Goetz C, Brandel JP, Lai EC, Wenning G, D'Olhaberriague L, Verny M, Chaudhuri KR, McKee A, Jellinger K, Bartko JJ, Mangone CA, Pearce RK. Accuracy of clinical criteria for the diagnosis of progressive supranuclear palsy (Steele-Richardson-Olszewski syndrome). Neurology. 1996 Apr;46(4):922-30. doi: 10.1212/wnl.46.4.922. PMID 8780065
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Min SW, Cho SH, Zhou Y, Schroeder S, Haroutunian V, Seeley WW, Huang EJ, Shen Y, Masliah E, Mukherjee C, Meyers D, Cole PA, Ott M, Gan L. Acetylation of tau inhibits its degradation and contributes to tauopathy. Neuron. 2010 Sep 23;67(6):953-66. doi: 10.1016/j.neuron.2010.08.044. PMID 20869593
- [Background] Randolph C, Tierney MC, Mohr E, Chase TN. The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): preliminary clinical validity. J Clin Exp Neuropsychol. 1998 Jun;20(3):310-9. doi: 10.1076/jcen.20.3.310.823. PMID 9845158
- [Background] Schneider LS, Olin JT, Doody RS, Clark CM, Morris JC, Reisberg B, Schmitt FA, Grundman M, Thomas RG, Ferris SH. Validity and reliability of the Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change. The Alzheimer's Disease Cooperative Study. Alzheimer Dis Assoc Disord. 1997;11 Suppl 2:S22-32. doi: 10.1097/00002093-199700112-00004. PMID 9236949
- [Background] Schrag A, Ben-Shlomo Y, Quinn NP. Prevalence of progressive supranuclear palsy and multiple system atrophy: a cross-sectional study. Lancet. 1999 Nov 20;354(9192):1771-5. doi: 10.1016/s0140-6736(99)04137-9. PMID 10577638
- [Background] Schrag A, Selai C, Quinn N, Lees A, Litvan I, Lang A, Poon Y, Bower J, Burn D, Hobart J. Measuring quality of life in PSP: the PSP-QoL. Neurology. 2006 Jul 11;67(1):39-44. doi: 10.1212/01.wnl.0000223826.84080.97. PMID 16832075
- [Background] Schwab RS and England Jr AC. 1969. Projection techniques for evaluating surgery in Parkinson's disease. In: Gilingham FJ and Donaldson IML, eds. Third symposium on Parkinson's disease. Edinburgh: E & S Livingstone Ltd. 152-157.
- [Background] STEELE JC, RICHARDSON JC, OLSZEWSKI J. PROGRESSIVE SUPRANUCLEAR PALSY. A HETEROGENEOUS DEGENERATION INVOLVING THE BRAIN STEM, BASAL GANGLIA AND CEREBELLUM WITH VERTICAL GAZE AND PSEUDOBULBAR PALSY, NUCHAL DYSTONIA AND DEMENTIA. Arch Neurol. 1964 Apr;10:333-59. doi: 10.1001/archneur.1964.00460160003001. No abstract available. PMID 14107684
- [Background] Strauss E, Sherman EMS, Spreen O. 2006. A compendium of neuropsychological tests: Administration, norms and commentary. 3rd ed. New York: Oxford University Press.
- [Background] Wenning GK, Litvan I, Jankovic J, Granata R, Mangone CA, McKee A, Poewe W, Jellinger K, Ray Chaudhuri K, D'Olhaberriague L, Pearce RK. Natural history and survival of 14 patients with corticobasal degeneration confirmed at postmortem examination. J Neurol Neurosurg Psychiatry. 1998 Feb;64(2):184-9. doi: 10.1136/jnnp.64.2.184. PMID 9489528
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Yoshiyama Y, Lee VM, Trojanowski JQ. Therapeutic strategies for tau mediated neurodegeneration. J Neurol Neurosurg Psychiatry. 2013 Jul;84(7):784-95. doi: 10.1136/jnnp-2012-303144. Epub 2012 Oct 20. PMID 23085937